CLINICAL TRIAL: NCT05351554
Title: A Randomized, Double-blind, Placebo-controlled, Phase 2a Study With an Open-label Cohort to Assess the Safety, Tolerability, and Efficacy of Namilumab in Subjects With Active Cardiac Sarcoidosis
Brief Title: A Study to Assess the Safety, Tolerability, and Efficacy of Namilumab in Participants With Active Cardiac Sarcoidosis
Acronym: RESOLVE-Heart
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor business decision not related to safety
Sponsor: Kinevant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KIN-1902-2002
Record Dates: First submitted 2022-04-04; First posted 2022-04-28 (Actual); Results first posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-02

CONDITIONS: Sarcoidosis, Cardiac
MeSH Terms: conditions — Sarcoidosis | interventions — namilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Namilumab (Experimental): A single participant received two doses of 150 milligrams (mg) of namilumab subcutaneously (SC) at baseline (Day 1) and on Day 15.
  Interventions: Drug: Namilumab

INTERVENTIONS:
Drug: Namilumab — Specified dose on specified days

SUMMARY:
A Randomized, Double-blind, Placebo-controlled, Study with an Open-label Cohort.

DETAILED DESCRIPTION:
Study was terminated after a single participant had received 2 doses.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age ≥18 years
* Able and willing to provide written informed consent, which includes compliance with study requirements and restrictions listed in the consent form
* History of documented sarcoidosis (must include histological confirmation, from any organ, in the subject's medical history or records)
* Meet Heart Rhythm Society Cardiac Sarcoid Diagnostic Criteria (modified)
* Female subjects must agree to use an approved highly effective birth control (BC) method
* Male subjects must agree to, and attest that, female partners of childbearing potential are using one of the allowed highly effective methods of contraception
* Body Mass Index (BMI) <40 kg/m2 at Screening.
* Vaccination for COVID-19 with completion of the primary series at least 2 weeks prior to randomization

Exclusion Criteria:

* Hospitalized for any respiratory or cardiac illness ≤30 days prior to Screening
* Known pulmonary hypertension requiring therapy
* Autoimmune disease other than sarcoidosis likely to require treatment during the subject's participation in this study
* Symptoms and/or signs of extracardiac sarcoidosis that are likely to warrant treatment in addition to that required for the subject's cardiac disease
* Estimated glomerular filtration rate (eGFR) ≤30 mL/min/1.73 m2 (Modification of Diet in Renal Disease [MDRD] equation) or requiring renal replacement therapy
* Hemoglobin ≤9.5 g/dL
* Participation in another interventional clinical trial within 6 months prior to Screening and throughout the duration of participation in this study
* Systolic blood pressure (SBP) <90 or >180 mm Hg; Diastolic blood pressure (DBP) <60 or >110 mm Hg at Screening
* Has documented laboratory-confirmed severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) infection as determined by polymerase chain reaction (PCR) or other approved clinical testing ≤3 months prior to randomization
* Significant valvular heart disease known or anticipated to require surgical repair or replacement during the subjects' participation in this study
* Female subjects who are pregnant or breastfeeding or intend to be, during the study
* History of severe allergic or anaphylactic reactions to therapeutic proteins or known sensitivity to namilumab or to its inactive components
* Any other acute or chronic medical condition, that in the judgment of the Investigator or Sponsor, may increase the risk associated with study participation or investigational product administration, or may interfere with the interpretation of study results, and would make the participant inappropriate for entry into this study

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-12-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Kinevant Study Site, Palo Alto, California
  - Kinevant Study Site, Denver, Colorado
  - Kinevant Study Site, New Haven, Connecticut
  - Kinevant Study Site, Gainesville, Florida
  - Kinevant Study Site, Iowa City, Iowa
  - Kinevant Study Site, Baltimore, Maryland
  - Kinevant Study Site, Boston, Massachusetts
  - Kinevant Study Site, Ann Arbor, Michigan
  - Kinevant Study Site, New York, New York
  - Kinevant Study Site, Cleveland, Ohio
  - Kinevant Study Site, Portland, Oregon
  - Kinevant Study Site, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The sponsor terminated the study for business reasons, not related to safety, after a single subject had received 2 doses. A separate cohort (Cohort A) was planned but did not enroll any participants.
Groups:
- Namilumab: A single participant received two doses of 150 mg (milligrams) of namilumab subcutaneously (SC) at baseline (Day 1) and on Day 15.
Period: Overall Study
Arm/Group | Namilumab
Started | 1
Received at Least 1 Dose of Study Drug | 1
Completed | 0
Not Completed | 1
Not completed — Study terminated by sponsor | 1

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least one dose of study drug.
Groups:
- Namilumab: A single participant received two doses of 150 mg of namilumab SC at baseline (Day 1) and on Day 15.
Arm/Group | Namilumab
Number analyzed (Participants) | 1
Age, Customized [Count of Participants; unit: Participants]
  50 - 70 years | 1
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male or Female | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), and AEs Leading to Discontinuation
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAEs were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to approximately 2 months
Population: The Safety Population included all randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Namilumab
Number analyzed (Participants) | 1
Participants
  AEs | 1
  SAEs | 0
  AEs leading to discontinuation | 0

2. Secondary Outcome: Number of Participants With Treatment-emergent Laboratory Abnormalities
Time Frame: Baseline up to approximately 2 months
Population: The Safety Population included all randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Namilumab
Number analyzed (Participants) | 1
Participants | 0

3. Secondary Outcome: Number of Participants With Treatment-emergent Vital Sign Abnormalities
Time Frame: Baseline up to approximately 2 months
Population: The Safety Population included all randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Namilumab
Number analyzed (Participants) | 1
Participants | 0

4. Secondary Outcome: Number of Participants With Treatment-emergent Electrocardiogram (ECG) Abnormalities
Time Frame: Baseline up to approximately 2 months
Population: The Safety Population included all randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Namilumab
Number analyzed (Participants) | 1
Participants | 0

5. Secondary Outcome: Mean Change From Baseline in Positron Emission Tomography (PET) Maximum Standardized Update Value (SUVmax)
Time Frame: Baseline up to approximately 2 months
Population: The study was terminated by the Sponsor due to a business decision (no safety concerns). The study participant did not consent to publishing his/her individual data. As there was only 1 participant in this study, no data are reported in order to protect and maintain participant privacy/confidentiality.
Arm/Group | Namilumab
Number analyzed (Participants) | 0

6. Secondary Outcome: Change From Baseline in PET Mean Standardized Update Value (SUVmean)
Time Frame: Baseline up to approximately 2 months
Population: as for outcome 5
Arm/Group | Namilumab
Number analyzed (Participants) | 0

7. Secondary Outcome: Mean Change From Baseline in Total Glycosylation
Time Frame: Baseline up to approximately 2 months
Population: as for outcome 5
Arm/Group | Namilumab
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Participants Hospitalized for Cardiac Events
Time Frame: Baseline up to approximately 2 months
Population: as for outcome 5
Arm/Group | Namilumab
Number analyzed (Participants) | 0

9. Secondary Outcome: Mean Change From Baseline in Left Ventricular Ejection Fraction (LVEF)
Time Frame: Baseline up to approximately 2 months
Population: as for outcome 5
Arm/Group | Namilumab
Number analyzed (Participants) | 0

10. Secondary Outcome: Mean Change From Baseline in Global Longitudinal Strain (GLS) on Transthoracic Echocardiogram (TTE)
Time Frame: Baseline up to approximately 2 months
Population: as for outcome 5
Arm/Group | Namilumab
Number analyzed (Participants) | 0

11. Secondary Outcome: Cumulative Oral Steroid Use
Time Frame: Baseline up to approximately 2 months
Population: as for outcome 5
Arm/Group | Namilumab
Number analyzed (Participants) | 0

12. Secondary Outcome: Modified Glucocorticoid Toxicity Index (mGTI)
Description: The mGTI is a composite measure of the changes in OCS toxicity measured at 3-month intervals across 11 domains and 23 items. For the purposes of this study, radiographic assessment of bone mineral density is not being performed; therefore, this item is not being assessed in the tool and the tool is termed "modified" for this study. The change in the total score is from -35 to +410 with the exclusion of bone mineral density, with minimum score representing least toxicity (better outcomes) and maximum score representing most toxicity (worse outcomes).
Time Frame: Baseline up to approximately 2 months
Population: as for outcome 5
Arm/Group | Namilumab
Number analyzed (Participants) | 0

13. Secondary Outcome: Mean Change From Baseline in Glycosylated Hemoglobin (HbA1C)
Time Frame: Baseline up to approximately 2 months
Population: as for outcome 5
Arm/Group | Namilumab
Number analyzed (Participants) | 0

14. Secondary Outcome: Number of Participants Requiring Rescue Therapy
Time Frame: Baseline up to approximately 2 months
Population: as for outcome 5
Arm/Group | Namilumab
Number analyzed (Participants) | 0

15. Secondary Outcome: Number of Participants Successfully Achieving Steroid Taper Without Requiring Rescue Therapy (Cohort A)
Time Frame: Baseline up to approximately 2 months
Population: 0 participants were enrolled in Cohort A.
Groups:
- Cohort A: Participants in Cohort A were to be randomized to either Namilumab or Placebo
Arm/Group | Cohort A
Number analyzed (Participants) | 0

16. Secondary Outcome: Mean Change From Baseline in King's Sarcoidosis Questionnaire (KSQ)
Description: The KSQ is a modular, multi-organ health status measure for participants with sarcoidosis for use in the clinic and the evaluation of therapies. The KSQ consists of 5 modules: General health status (10 items), Lung (6 items), Medication (3 items), Skin (3 items), and Eye (7 items). Results are given as a number between 1-100 with higher numbers indicating better health.
Time Frame: Baseline up to approximately 2 months
Population: as for outcome 5
Arm/Group | Namilumab
Number analyzed (Participants) | 0

17. Secondary Outcome: Change From Baseline in Fatigue Assessment Scale (FAS)
Description: The FAS is a 10-item self-reported fatigue questionnaire. Participants indicate their responses on a 5-point scale (from 1 never to 5 always). Total scores on the FAS can therefore range from 10 to 50, with high scores indicating more fatigue and worse outcomes.
Time Frame: Baseline up to approximately 2 months
Population: as for outcome 5
Arm/Group | Namilumab
Number analyzed (Participants) | 0

18. Secondary Outcome: Change From Baseline in Subject Global Assessment (SGA)
Description: The SGA is a participant reported outcome instrument used to assess their overall perception of the frequency and severity of sarcoid symptoms. The SGA is a 5-point Likert scale; the participant rates how he/she feels regarding their sarcoidosis in the previous 2 weeks prior to the study visit based on the frequency and severity of their symptoms. Scores range from 1 to 5 with lower scores representing better outcomes.
Time Frame: Baseline up to approximately 2 months
Population: as for outcome 5
Arm/Group | Namilumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to approximately 2 months
Groups:
- Namilumab: Participant received two doses of 150 mg of namilumab SC at baseline (Day 1) and on Day 15.
Arm/Group | Namilumab
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Namilumab (N=1)
Rash (Skin and subcutaneous tissue disorders) | 1
Headache (Nervous system disorders) | 1
Injection site papule (General disorders) | 1

LIMITATIONS AND CAVEATS:
The sponsor terminated the study for business reasons, not related to safety, after a single participant had received 2 doses. No efficacy analyses were performed and no conclusions can be drawn due to the limited data available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/54/NCT05351554/Prot_SAP_000.pdf